CLINICAL TRIAL: NCT04549896
Title: Interest of Coronary CT Scan Before Complex Chronic Total Occlusion (CTO) Percutaneous Coronary Intervention (PCI).
Brief Title: Computed Tomography Scan in Complex Chronic Total Occlusion Percutaneous Coronary Intervention;
Acronym: CTS-C-CTOPCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTS-C-CTOPCI
Record Dates: First submitted 2020-07-29; First posted 2020-09-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Total Occlusion of Coronary Artery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT scan (Experimental): CT scan with a last generation 256 slice machine of occluded coronary artery before CTO PCI
  Interventions: Procedure: CT scan
- Control (Active Comparator): No CT scan before CTO PCI
  Interventions: Procedure: No CT scan

INTERVENTIONS:
Procedure: CT scan — Surgeon will perform a CT scan before the surgery procedure (CTO PCI) in order to increase the success rate of the surgery.
  Arms: CT scan
Procedure: No CT scan — The surgery procedure (CTO PCI) will be performed following the standard of care, meaning that the surgeon will not perform a CT scan before the surgery procedure.
  Arms: Control

SUMMARY:
The chronic total occlusion of a coronary artery is the most frequent cardiac disease in the developped countries. The percutaneous coronary intervention is one of the existing treatments. This procedure is long, expensive and uses a lot of contrast medium and X ray. With this study, the investigators want to adress the impact of CT scan performed before the surgical procedure. A better knowledge of the patient's anatomy could lead to a better success rate of the operation, with a lower radiation, lower contrast injection, and a faster and more cost-efficient procedure.

DETAILED DESCRIPTION:
A chronic total occlusion (CTO) is the complete obstruction of a coronary artery that has been established from more than 3 months with TIMI (Thrombolysis in Myocardial Infarction) 0 flow. This is a frequent pathology, demonstrated in 20% of patients studied with a coronary angiography. The patients affected by an isolated CTO or by a multi-vascular coronary disease with one or more CTO are an heterogenous population in relation to age, co-morbidity, risk factors.

The treatment of this disease is medical, interventional or surgical. The interventional option is often the first choice in case of symptoms or ischemia associated with viability of the myocardial wall, originally perfused by the occluded segment. Medical treatment is often not enough to reduce symptoms and to improve quality of life. Surgery is very invasive, especially for patients with mono-vascular disease, not always possible, especially in case of distal diffuse disease or heavy co-morbidity.

The Percutaneous Coronary Intervention (PCI) is a good option thanks to the improvement of materials and recanalization techniques (anterograde, retrograde and dissection re-entry). However, the procedure is often long, expensive, using a lot of contrast medium and X ray.

At the diagnosis stage of a CTO, the Japan Chronic Total Occlusion (J-CTO) score defines the complexity of the procedure : 0 easy, 1 intermediate, 2 hard, ≥ 3 very hard. The score is actually calculated with the angiography data after evaluation of the occlusion's proximal cap shape, presence of calcifications in the occluded segment, tortuosity of the occluded segment and length of the occlusion.

In addition to the angiography data, a CT scan of coronary artery can be performed as part of Standard of Care. In the study's coordinating center, more than 2000 CT scans are performed by the team of interventional cardiologists. Data generated from last generation CT scan are then interpreted to extrapolate informations about the occluded segment, the occluded artery and the contralateral artery.

CT scan is able to identify very well the calcium distribution in the occluded segment/artery, the true length of the occlusion, bends, collateral branches, distal vessel anatomy, coronary path and more, solving ambiguity of proximal cap and showing the shape of the distal cap. Thanks to this investigation, the investigators can better evaluate the J-CTO score and the CT Rector score. The CT Rector score is helping to grade the CTO difficulty before the PCI by predicting time-efficient guidewire crossing. The investigators can calculate the calcium score of the occluded artery to detect a critical value for the success of CTO PCI. The best strategy with appropriate material can then be chosen for the procedure PCI.

In this study, the investigators would like to demonstrate the interest in performing a CT scan as a part of the pathology diagnosis before the PCI in more complex occlusions (J-CTO score ≥ 2). The investigators think that the CT scan, with a last generation GE Revolution 256 slice machine, is actually the best method to evaluate the J-CTO score, the CT Rector score and to obtain other important information like anatomical position of the occluded artery and presence of side branches in the occluded segment.

A better evaluation of J-CTO score and complex anatomy will then allow the selection of the best technique for the procedure with probably a better success rate, lower radiation, lower contrast injection, and a faster and more cost-efficient procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old and ≤ 90 years old,
2. BMI ≤ 40 kg/m²,
3. Dated and signed informed consent, before any study-related procedures
4. Ability to understand and comply with the study procedures,
5. Affiliate or recipient of a social security scheme,
6. Coronary artery chronic total occlusion (TIMI 0 flow from > 3 months) associated with myocardial viability (intended like normokinetic/hypokinetic wall motion or instrumental data in favor of viability) associated with ≥ CCS2 angina or ≥ NHYA2 dyspnea or documented ischemia or ejection fraction <50%.
7. Coronary angiography J-CTO score ≥ 2 (complex cases)

Exclusion Criteria:

1. Pregnant or breastfeeding woman,
2. Adults patients protected by law,
3. Very frequent and irregular cardiac rhythm (>100/min.),
4. More than one CTO to be treated by PCI,
5. Coronary angiography J-CTO (Japan Chronic Total Occlusion) score 0/1
6. Hemodynamic instability,
7. Anemia < 9g/dl,
8. Gastrointestinal bleeding,
9. Thrombocytopenia with < 50 000/mm3 platelets count,
10. Severe valvular disease associated
11. CT-Scan performed as part of the standard of care pathology diagnosis, before the inclusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful CTO PCI procedure in both groups | Immediately after surgery.
  TIMI 3 flow restoration and residual stenosis < 30%, by wire crossing in less than (≤) 60 minutes guidewire manipulation. TIMI flow and residual stenosis will be evaluated by a pool of 2 cardiologists not involved in the procedure and blinded regarding the randomized group.

SECONDARY OUTCOMES:
Total time of CTO PCI procedure | Immediately after surgery.
  Duration of the surgery procedure given in minutes.
Rate of CTO PCI complications | 6 months starting from the date of the surgery.
  Death, coronary perforation with cardiac tamponade requiring pericardiocentesis, myocardial infarction (if elevation of troponin/CK associated with change in electrocardiogram), stroke, major bleeding with lost of hemoglobin > 3g/dl.
Radiation level used during the CTO PCI procedure | Immediately after surgery.
  Quantity of radiation used during the PCI (airKerma in Gy, DAP mGycm², fluoroscopy time in minutes).
Volume of iodine contrast medium used for the CTO PCI procedure | Immediately after surgery.
  Quantity of iodine contrast medium used during the PCI (given in milliliters).
Cost of the the CTO PCI procedure | Immediately after surgery.
  Total cost of the surgery procedure (given in euros).
Creatinine level before discharge | 24 hours after surgery
  This endpoint summarizes the renal adverse events in both groups. A baseline creatinine level is always known before the coronary angiography that initializes the diagnostic and therapeutic pathway.
Safety assessed with Adverse Events reporting | 6 months starting from the date of the surgery.
  Any adverse events will be reported (like contrast allergic reaction). Their relationship with the CT scan or PCI procedure will also be reported.
Angina and dyspnea | 6 months starting from the date of the inclusion.
  Symptoms (angina CCS class / dyspnea NYHA (New York Heart Association) class) will be collected at the CTO PCI visit and EOS visit.
Major Adverse Cardiac Events | 6 months starting the date of the inclusion.
  Major Adverse Cardiac Events (MACE: myocardial infarction, cardiovascular death, revascularization, stroke) will be collected at the CTO PCI visit and EOS visit.
renal failure collection | 6 months starting the date of the inclusion.
  Renal failure will be collected at the CTO PCI visit and EOS visit.
Troponin measure | Baseline.
  Levels of troponin will be reported.
CK measure | Baseline.
  Levels of CK will be reported.
Creatinine measure | Baseline.
  Levels of creatinine will be reported.
clearance of creatinine measure | Baseline.
  Levels of the clearance of creatinine will be reported.
Hemoglobin measure | Baseline.
  Levels of hemoglobin will be reported.
Troponin measure | 24 hours after surgery
  Levels of troponin will be reported after the PCI at the CTO PCI visit.
CK measure | 24 hours after surgery
  Levels of CK will be reported after the PCI at the CTO PCI visit.
Creatinine measure | 24 hours after surgery
  Levels of creatinine will be reported after the PCI at the CTO PCI visit.
clearance of creatinine measure | 24 hours after surgery
  Levels of the clearance of creatinine will be reported after the PCI at the CTO PCI visit.
Hemoglobin measure | 24 hours after surgery
  Levels of hemoglobin will be reported after the PCI at the CTO PCI visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique Les Fleurs, Ollioules, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesebro JH, Knatterud G, Roberts R, Borer J, Cohen LS, Dalen J, Dodge HT, Francis CK, Hillis D, Ludbrook P, et al. Thrombolysis in Myocardial Infarction (TIMI) Trial, Phase I: A comparison between intravenous tissue plasminogen activator and intravenous streptokinase. Clinical findings through hospital discharge. Circulation. 1987 Jul;76(1):142-54. doi: 10.1161/01.cir.76.1.142. PMID 3109764
- [Background] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Background] Morino Y, Abe M, Morimoto T, Kimura T, Hayashi Y, Muramatsu T, Ochiai M, Noguchi Y, Kato K, Shibata Y, Hiasa Y, Doi O, Yamashita T, Hinohara T, Tanaka H, Mitsudo K; J-CTO Registry Investigators. Predicting successful guidewire crossing through chronic total occlusion of native coronary lesions within 30 minutes: the J-CTO (Multicenter CTO Registry in Japan) score as a difficulty grading and time assessment tool. JACC Cardiovasc Interv. 2011 Feb;4(2):213-21. doi: 10.1016/j.jcin.2010.09.024. PMID 21349461
- [Background] Rolf A, Werner GS, Schuhback A, Rixe J, Mollmann H, Nef HM, Gundermann C, Liebetrau C, Krombach GA, Hamm CW, Achenbach S. Preprocedural coronary CT angiography significantly improves success rates of PCI for chronic total occlusion. Int J Cardiovasc Imaging. 2013 Dec;29(8):1819-27. doi: 10.1007/s10554-013-0258-y. Epub 2013 Jun 23. PMID 23793727
- [Background] Yu CW, Lee HJ, Suh J, Lee NH, Park SM, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee SH, Choe YH, Kim SM, Choi JH. Coronary Computed Tomography Angiography Predicts Guidewire Crossing and Success of Percutaneous Intervention for Chronic Total Occlusion: Korean Multicenter CTO CT Registry Score as a Tool for Assessing Difficulty in Chronic Total Occlusion Percutaneous Coronary Intervention. Circ Cardiovasc Imaging. 2017 Apr;10(4):e005800. doi: 10.1161/CIRCIMAGING.116.005800. PMID 28389507
- [Background] Singh S, Singh N, Gulati GS, Ramakrishnan S, Kumar G, Sharma S, Bahl VK. Dual-Source Computed Tomography for Chronic Total Occlusion of Coronary Arteries. Catheter Cardiovasc Interv. 2016 Oct;88(4):E117-E125. doi: 10.1002/ccd.25516. Epub 2014 May 27. PMID 24740894
- [Background] Ghoshhajra BB, Takx RAP, Stone LL, Girard EE, Brilakis ES, Lombardi WL, Yeh RW, Jaffer FA. Real-time fusion of coronary CT angiography with x-ray fluoroscopy during chronic total occlusion PCI. Eur Radiol. 2017 Jun;27(6):2464-2473. doi: 10.1007/s00330-016-4599-5. Epub 2016 Sep 23. PMID 27663227
- [Background] Li Y, Xu N, Zhang J, Li M, Lu Z, Wei M, Lu B, Zhang Y. Procedural success of CTO recanalization: Comparison of the J-CTO score determined by coronary CT angiography to invasive angiography. J Cardiovasc Comput Tomogr. 2015 Nov-Dec;9(6):578-84. doi: 10.1016/j.jcct.2015.07.005. Epub 2015 Jul 23. PMID 26232276
- [Background] Opolski MP, Achenbach S. CT Angiography for Revascularization of CTO: Crossing the Borders of Diagnosis and Treatment. JACC Cardiovasc Imaging. 2015 Jul;8(7):846-58. doi: 10.1016/j.jcmg.2015.05.001. PMID 26183556
- [Background] Chen Y, Lu B, Hou ZH, Gao Y, Yu FF, Yin WH, Wang ZQ. Predicting successful percutaneous coronary intervention in patients with chronic total occlusion: the incremental value of a novel morphological parameter assessed by computed tomography. Int J Cardiovasc Imaging. 2015 Aug;31(6):1263-9. doi: 10.1007/s10554-015-0679-x. Epub 2015 May 17. PMID 25982175
- [Background] Opolski MP, Achenbach S, Schuhback A, Rolf A, Mollmann H, Nef H, Rixe J, Renker M, Witkowski A, Kepka C, Walther C, Schlundt C, Debski A, Jakubczyk M, Hamm CW. Coronary computed tomographic prediction rule for time-efficient guidewire crossing through chronic total occlusion: insights from the CT-RECTOR multicenter registry (Computed Tomography Registry of Chronic Total Occlusion Revascularization). JACC Cardiovasc Interv. 2015 Feb;8(2):257-267. doi: 10.1016/j.jcin.2014.07.031. PMID 25700748
- [Background] Takimura H, Muramatsu T, Tsukahara R. CT coronary angiography-guided percutaneous coronary intervention for chronic total occlusion combined with retrograde approach. J Invasive Cardiol. 2012 Jan;24(1):E5-9. PMID 22210595
- [Background] Rodriguez-Granillo GA, Rosales MA, Llaurado C, Ivanc TB, Rodriguez AE. Guidance of percutaneous coronary interventions by multidetector row computed tomography coronary angiography. EuroIntervention. 2011 Jan;6(6):773-8. doi: 10.4244/EIJV6I6A131. PMID 21205604
- [Background] Tajti P, Karmpaliotis D, Alaswad K, Jaffer FA, Yeh RW, Patel M, Mahmud E, Choi JW, Burke MN, Doing AH, Dattilo P, Toma C, Smith AJC, Uretsky B, Holper E, Wyman RM, Kandzari DE, Garcia S, Krestyaninov O, Khelimskii D, Koutouzis M, Tsiafoutis I, Moses JW, Lembo NJ, Parikh M, Kirtane AJ, Ali ZA, Doshi D, Rangan BV, Ungi I, Banerjee S, Brilakis ES. The Hybrid Approach to Chronic Total Occlusion Percutaneous Coronary Intervention: Update From the PROGRESS CTO Registry. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1325-1335. doi: 10.1016/j.jcin.2018.02.036. Epub 2018 Apr 26. PMID 29706508
- [Background] Maeremans J, Walsh S, Knaapen P, Spratt JC, Avran A, Hanratty CG, Faurie B, Agostoni P, Bressollette E, Kayaert P, Bagnall AJ, Egred M, Smith D, Chase A, McEntegart MB, Smith WH, Harcombe A, Kelly P, Irving J, Smith EJ, Strange JW, Dens J. The Hybrid Algorithm for Treating Chronic Total Occlusions in Europe: The RECHARGE Registry. J Am Coll Cardiol. 2016 Nov 1;68(18):1958-1970. doi: 10.1016/j.jacc.2016.08.034. PMID 27788851
- [Background] Hunt CH, Hartman RP, Hesley GK. Frequency and severity of adverse effects of iodinated and gadolinium contrast materials: retrospective review of 456,930 doses. AJR Am J Roentgenol. 2009 Oct;193(4):1124-7. doi: 10.2214/AJR.09.2520. PMID 19770337
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Galassi AR, Sianos G, Werner GS, Escaned J, Tomasello SD, Boukhris M, Castaing M, Buttner JH, Bufe A, Kalnins A, Spratt JC, Garbo R, Hildick-Smith D, Elhadad S, Gagnor A, Lauer B, Bryniarski L, Christiansen EH, Thuesen L, Meyer-Gessner M, Goktekin O, Carlino M, Louvard Y, Lefevre T, Lismanis A, Gelev VL, Serra A, Marza F, Di Mario C, Reifart N; Euro CTO Club. Retrograde Recanalization of Chronic Total Occlusions in Europe: Procedural, In-Hospital, and Long-Term Outcomes From the Multicenter ERCTO Registry. J Am Coll Cardiol. 2015 Jun 9;65(22):2388-400. doi: 10.1016/j.jacc.2015.03.566. PMID 26046732
- [Background] Patel VG, Brayton KM, Tamayo A, Mogabgab O, Michael TT, Lo N, Alomar M, Shorrock D, Cipher D, Abdullah S, Banerjee S, Brilakis ES. Angiographic success and procedural complications in patients undergoing percutaneous coronary chronic total occlusion interventions: a weighted meta-analysis of 18,061 patients from 65 studies. JACC Cardiovasc Interv. 2013 Feb;6(2):128-36. doi: 10.1016/j.jcin.2012.10.011. Epub 2013 Jan 23. PMID 23352817
- [Background] Hannan EL, Zhong Y, Jacobs AK, Stamato NJ, Berger PB, Walford G, Sharma S, Venditti FJ, King SB 3rd. Patients With Chronic Total Occlusions Undergoing Percutaneous Coronary Interventions: Characteristics, Success, and Outcomes. Circ Cardiovasc Interv. 2016 May;9(5):e003586. doi: 10.1161/CIRCINTERVENTIONS.116.003586. PMID 27162216
- [Background] Brilakis ES, Banerjee S, Karmpaliotis D, Lombardi WL, Tsai TT, Shunk KA, Kennedy KF, Spertus JA, Holmes DR Jr, Grantham JA. Procedural outcomes of chronic total occlusion percutaneous coronary intervention: a report from the NCDR (National Cardiovascular Data Registry). JACC Cardiovasc Interv. 2015 Feb;8(2):245-253. doi: 10.1016/j.jcin.2014.08.014. PMID 25700746
- [Derived] La Scala E, Peyre JP, Maupas E; ReSurg; CT-CTO PCI Study Group. Effect of preoperative coronary CT for planning of percutaneous coronary intervention for complex chronic total occlusion (CTS-C-CTOPCI): study protocol for an open-label randomised controlled trial. Trials. 2023 Aug 29;24(1):560. doi: 10.1186/s13063-023-07458-y. PMID 37644573